CLINICAL TRIAL: NCT04032509
Title: A Prospective Clinical Study of Biomarkers of Mild Traumatic BRAIN Injury
Brief Title: A Study of Biomarkers of Mild Traumatic BRAIN Injury
Acronym: BRAINI
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.176; 2019-A01525-52 (Other: ID RCB)
Record Dates: First submitted 2019-07-15; First posted 2019-07-25 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2020-08

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild TBI: Mild TBI (GCS 13-15 on admission) within 12 hours after injury
  Interventions: Other: 2 x 5 mL blood sample

INTERVENTIONS:
Other: 2 x 5 mL blood sample — 2 x 5 mL blood sample to determine the performance of the automated VIDAS BTI platform in assessing serum concentrations of GFAP and UCH-L1 to rule out the need for a CT-scan after mTBI.

SUMMARY:
Patients with mild traumatic brain injury (mTBI) represent a burden of patients admitted to the emergency department. According to the guidelines, a cerebral CT scan is indicated after mTBI according to the specific conditions. However, variability exists regarding the respect of these CT scan indications, and less than 10% of patients will have visible brain lesions on CT scan. Recently, serum Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase-L1 (UCH-L1) biomarkers have shown ability to differentiate normal and abnormal CT scan findings after mTBI. These encouraging results prompted us to launch a prospective study using automated and quick measurements of GFAP and UCH-L1 biomarkers to validate these findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old (France)
* Mild TBI (GCS 13-15 on admission) within 12 hours after injury
* Indication of brain CT scan:

  * neurological focal deficit
  * anterograde amnesia
  * Glasgow coma scale score <15 after 2 hours post-TBI
  * suspicion of vault depression fracture
  * fracture of the basal skull
  * persisting nausea, vomiting or headache
  * post-TBI seizures
  * Pre-injury treatment with antithrombotic drugs
  * Loss of consciousness or amnesia with age >65 years, fall >1m or hit pedestrian
  * Other condition requiring CT scan according to the in-charge physician.

Exclusion Criteria:

* GCS 3-12 on admission
* Time of injury unknown
* Time to injury exceeding 12 hours
* Primary admission for non-traumatic neurological disorder (e.g., stroke, spontaneous intracranial hematoma)
* Penetrating head trauma
* Patient with mechanical ventilation
* Pre-injury neurological disorder affecting the assessment of neurological outcome: dementia, Parkinson's disease, multiple sclerosis, seizure disorder, brain tumor, and history of neurosurgery, stroke or transient ischemic attack (TIA) within the last 30 days
* Venipuncture not feasible
* No realization of brain CT-scan
* Subject under judiciary control
* Pregnant or breastfeeding woman
* Subject in exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1600 patients: 1300 patients in France and 300 patients in Spain
Sampling Method: Probability Sample
Enrollment: 1501 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Performance of the VIDAS-BTI assay in terms of sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and their corresponding lower limit of 95% confidence interval by comparison with brain CT scan findings. | 12 hours post Traumatic Brain Injury (TBI)
  2 x 5mL blood sample

SECONDARY OUTCOMES:
Determination of the added value of the two biomarkers measurements to Transcranial Doppler (TCD) performed on admission to detect patients at risk of neurological worsening and patients allowed for a safe return home | Admission
  TCD measures at admission
Determination of the added value of the two biomarkers measurements to Transcranial Doppler (TCD) performed on admission to detect patients at risk of neurological worsening and patients allowed for a safe return home | 7 days after traumatic brain injury (TBI)
  Neurological status at 1 week after TBI
Determination of the added value of the two biomarkers measurements to Transcranial Doppler (TCD) performed on admission to detect patients at risk of neurological worsening and patients allowed for a safe return home | 7 days after traumatic brain injury (TBI)
  Quality of life after brain injury (QOLIBRI) Questionnaire
Determination the potential of the two biomarkers in predicting neurological outcome | 3 month after TBI
  Extended Glasgow Outcome Scale (GOSE)
Determination of the potential of the two biomarkers in predicting neurological outcome | 3 month after TBI
  Quality of life after brain injury (QOLIBRI) Questionnaire)
Determination of the potential of the two biomarkers in predicting neurological outcome | 3 month after TBI
  EuroQuol 5 dimensions 5 level questionnaire (EQ-5D-5L)
Determination of the potential of the two biomarkers in predicting neurological outcome | 3 month after TBI
  Rivermead Post-concussion symptoms Questionnaire (RPQ)

CONTACTS AND LOCATIONS:
Locations (16):
- France (12):
  - Centre Hospitalier Annecy Genevois, Annecy
  - CHU Bordeaux, Bordeaux
  - CHU Dijon, Dijon
  - CHU Grenoble Alpes, Grenoble
  - Hopital Edouard HERRIOT - HCL, Lyon
  - Hopital Lyon Sud HCL, Lyon
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - Hôpital Nord Ouest de Villefranche sur Saône, Villefranche-sur-Saône
- Spain (4):
  - Hospital de La Princesa, Madrid
  - Hospital del Tajo, Madrid
  - Hospital Gregorio Maranon, Madrid
  - Hospital Universitario de 12 Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lagares A, de la Cruz J, Terrisse H, Mejan O, Pavlov V, Vermorel C, Payen JF; of the BRAINI participants and investigators. An automated blood test for glial fibrillary acidic protein (GFAP) and ubiquitin carboxy-terminal hydrolase L1 (UCH-L1) to predict the absence of intracranial lesions on head CT in adult patients with mild traumatic brain injury: BRAINI, a multicentre observational study in Europe. EBioMedicine. 2024 Dec;110:105477. doi: 10.1016/j.ebiom.2024.105477. Epub 2024 Nov 29. PMID 39612652
- [Derived] Richard M, Lagares A, Bondanese V, de la Cruz J, Mejan O, Pavlov V, Payen JF; BRAINI investigators. Study protocol for investigating the performance of an automated blood test measuring GFAP and UCH-L1 in a prospective observational cohort of patients with mild traumatic brain injury: European BRAINI study. BMJ Open. 2021 Feb 25;11(2):e043635. doi: 10.1136/bmjopen-2020-043635. PMID 33632753